CLINICAL TRIAL: NCT03611517
Title: SPARC Study: A Nurse-led Sexual Rehabilitation Programme for Women With Gynaecological Cancers Receiving Radiotherapy: a Randomized Multicentre Trial
Brief Title: Sexual Rehabilitation Programme After Radiotherapy for Gynaecological Cancer
Acronym: SPARC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Leiden University Medical Center (Other)
Collaborators: Dutch Cancer Society (Other)
Responsible Party: Principal Investigator, MMterKuile, PhD, clinical psychologist, associate professor, Leiden University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P17.317; 10674 (Other Grant/Funding Number: KWF Kankerbestrijding); NL62767.058.17 (Other: CCMO)
Record Dates: First submitted 2018-05-29; First posted 2018-08-02 (Actual); Last update posted 2020-02-24 (Actual); Status verified 2020-02

CONDITIONS: Endometrial Cancer; Cervical Cancer; Vaginal Cancer; Gynecologic Cancer
Keywords: Endometrial cancer; Cervical cancer; Vaginal cancer; sexuality; sexual problems; dilator; radiotherapy; gynaecological cancer; sexual rehabilitation programme
MeSH Terms: conditions — Endometrial Neoplasms; Uterine Cervical Neoplasms; Vaginal Neoplasms; Sexuality

STUDY DESIGN:
Intervention Model Description: After signed informed consent, women complete the baseline questionnaire. After completion of the baseline questionnaire and before the end of RT, patients will be randomized to either the intervention group or the control group. The control group receives care as usual. The intervention group receives the nurse-led sexual rehabilitation intervention. All patients have follow-up appointments with their radiation-oncologist (or gynecologic oncologist) at 1, 3, 6 and 12 months post RT. For the intervention group, the sexual rehabilitation intervention sessions with the nurse will be planned immediately following the appointment with the radiation-oncologist. Women in the intervention group who are treated with RTBT receive an extra session 2 months after the end of radiotherapy. All patients are asked to complete questionnaires at baseline, and 1, 3, 6, and 12 months after completion of RT.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sexual rehabilitation programme (Experimental): The intervention exists of a nurse-led sexual rehabilitation programme, which is provided in addition to the care as usual. The intervention consists of four one-hour sessions at 1 month, 3, 6, and 12 months after RT. Women treated with RTBT will receive an additional appointment with the nurse (2 months after RTBT). Furthermore, the latter group receives a vaginal dilator set.
  Interventions: Behavioral: Sexual rehabilitation programme
- Care as usual (No Intervention): The control group receives the optimal care as usual, according to each participating hospital's guidelines. Additionally, all patients receive an information booklet including information concerning sexuality after RT for GC. Patients who underwent RTBT also receive a vaginal dilator set.

INTERVENTIONS:
Behavioral: Sexual rehabilitation programme — The intervention consists of 4 patient/couple sessions (each max. 60 minutes) scheduled at 1, 3, 6 and 12 months post-RT. Patients treated with RTBT have an additional session 2 months post RT. If preferred, one extra session of 30 minutes can be scheduled between 6 and 12 months after RT. The intervention includes (1) education on the specific cancer diagnosis and treatment, (2) education on the importance of regular dilation for prevention of vaginal stenosis (if indicated), (3) discussing and resolving potential fears and experienced barriers to performing vaginal dilation (if indicated) and sexual activity,(4) promoting couples' mutual coping and support processes and (5) specific sexual therapy techniques to address sexual and body image concerns.
  Arms: Sexual rehabilitation programme

SUMMARY:
The aim of this randomized controlled trial is to demonstrate that a nurse-led sexual rehabilitation intervention significantly improves sexual recovery and functioning among gynaecological cancer (GC) patients treated with radiotherapy (RT), compared with usual care (i.e., oral information by a nurse or doctor and written information).

Women with GC (n=220) who receive RT in one of the participating Dutch GC centres (n=9) will be randomized to either the sexual rehabilitation intervention (n= 110) or usual care (n= 110), stratified for combined RTBT vs. RT alone, and for having a partner (yes/no). Women are eligible for participation if they: have been diagnosed with either cervical, endometrial, or vaginal cancer; are treated with radiotherapy; are 18 years or older; and wish to retain their sexual activity on the short or long term.

The intervention consists of four one-hour sessions at 1 month, 3, 6, and 12 months after RT. Women who received RTBT will receive an additional appointment with the nurse (2 months after RTBT) to promote regular use of vaginal dilators in order to prevent stenosis. Participants are requested to complete questionnaires at baseline and at 1, 3, 6, and 12 months post-RT.

The primary endpoint is sexual functioning at 12 months. Secondary endpoints include vaginal symptoms and body concerns, fear of coital and non-coital sexual activity, sexual distress, treatment-related distress, generic health-related quality of life, psychological distress, and relationship dissatisfaction.

Hypothesis: The investigators expect women who receive the nurse-led sexual rehabilitation programme to report a greater improvement in sexual functioning from immediate post-radiotherapy to 1 year post-radiotherapy than women in the control group.

DETAILED DESCRIPTION:
The primary objective of this randomized controlled trial is to evaluate if the nurse-led sexual rehabilitation intervention improves sexual recovery and functioning in patients with gynaecological cancers (GC) who are treated with either external pelvic radiotherapy only (i.e., RT) or external pelvic radiotherapy combined with brachytherapy (i.e., RTBT) compared with usual care (Q1).

The secondary objective is to evaluate if the nurse-led sexual rehabilitation program decreases vaginal symptoms and body image concerns, fear of (non-)coital sexual activity, treatment-related distress, psychological and sexual distress, and vaginal physical symptoms (assessed during physical examination by the radiation oncologist), and improves/increases generic-related health related quality of life related to gynaecological cancer, relationship satisfaction, and frequency of dilator use, (Q2); to evaluate the cost-effectiveness of the intervention (Q3); and to evaluate whether an improvement in sexual functioning is moderated by treatment characteristics and pre-treatment patient characteristics, such as age or sexual functioning, and mediated by reduction of vaginal symptoms (and by regular use of dilators in women treated with RTBT) (Q4).

ELIGIBILITY:
Inclusion Criteria:

* being diagnosed with on of the following gynaecological cancers: cervical cancer, endometrial cancer or vaginal cancer
* 18 years or older
* receiving radiotherapy for gynaecological cancer (RT/RTBT)
* wish to retain sexual activity in the short- or long-term.

Exclusion Criteria:

* being unavailable for follow-up
* having insufficient knowlegde of the Dutch language
* having a psychiatric disorder (e.g. major affective disorder, psychotic disorder, substance abuse disorder (i.e., alcohol, drugs), or posttraumatic stress disorder resulting from abuse in the pelvic floor and/or genitals (e.g., sexual abuse)).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2018-08-07 (Actual); Primary Completion 2022-07 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
Change from 1 month in Sexual functioning at 12 months post RT/RTBT | 12 months
  The primary outcome measure is sexual functioning and will be assessed with the Dutch version of the 19-item Female Sexual Function Index (FSFI) questionnaire. The FSFI consists of 6 subscales measuring sexual desire (scoring range: 0.6 - 6.0), arousal (scoring range: 0 - 6.0), lubrication (scoring range: 0 - 6.0), orgasm (scoring range: 0 - 6.0), satisfaction (scoring range: 0.8 - 6.0), and pain (scoring range: 0 - 6.0). The scores of the questions are added per subscale, after which they are multiplied by a factor depending on the subscale ( sexual desire: 0.6; arousal: 0.3; lubrication: 0.3; orgasm: 0.4; satisfaction: 0.4; pain: 0.4) to give them a subscale score. By adding all 6 subscales together, the total score of the FSFI is obtained. The total score reflects overall sexual functioning (scoring range: 2.0 - 36.0). Higher scores indicate better sexual functioning. (measured at 1, 3, 6, 12 months post RT/RTBT and retrospectively (sexual functioning before diagnosis) at baseline

SECONDARY OUTCOMES:
Changes from 1 month in Vaginal symptoms and body image concerns at 12 months post RT/RTBT | 12 months
  Vaginal symptoms and body image concerns will be assessed with the Quality-of-Life Questionnaire (QLQ) Cervical Cancer Module (CX24) and Endometrial Cancer Module (EN24) of the Dutch version of the European Organization for Research and Treatment of Cancer (EORTC; EORTC-QLQ-CX24, EORTC-QLQ-EN24). The EORTC-QLQ-CX24 consists of 9 subscales: symptom experience (scoring range 11 - 44), lymphoedema (scoring range: 1-4), peripheral neuropathy (scoring range: 1-4), menopausal symptoms (scoring range: 1-4), sexual worry (scoring range: 1-4), body image (scoring range: 3-12), sexual activity (scoring range: 1-4), sexual enjoyment (scoring range: 1-4), sexual/vaginal functioning (scoring range: 4-16). Items 34, 38, 39, 40, 42, and 49 of the EORTC-QLQ-EN24 will be assessed (item range: 3). Lower scores indicate better sexual/vaginal functioning and lower body image concerns and relevant subscales. (measured at 1, 3, 6, 12 months post RT/RTBT).
Change from 1 month in Fear of coital and non-coital sexual activity at 12 months post RT/RTBT | 12 months
  Fear of coital and non-coital sexual activity will be assessed with the 8-item Fear of Sexuality Questionnaire (FSQ). The FSQ consist of 2 subscales: fear of non-coital sexual activity (scoring range: 5-25), and fear of coitus (scoring range:3-15). A higher score indicates more fear. (measured at 1, 3, 6, 12 months post RT/RTBT).
Change from 1 month in Level of sexual distress at 12 months post RT/RTBT | 12 months
  The level of sexual distress is assessed with the 12-item (scoring range: 0-48)Female Sexual Distress Scale (FSDS). Higher scores indicate more sexual dissatisfaction/distress. (measured at 1, 3, 6, 12 months post RT/RTBT and at baseline (retrospectively) concerning sexual functioning before diagnosis).
Change from 1 month in Treatment related distress at 12 months post RT/RTBT | 12 months
  Treatment related distress is assessed with Dutch version of the 15-items Impact of Event Scale-revised (IES-R; in Dutch Schokverwerkingslijst (SVL)). The total scores on the IES-R have a possible range of 0-75, with higher scores indicating a greater frequency of intrusive thoughts and attempts at avoidance. Subscale scores can also be computed for the 7 intrusion items (scoring range: 0-35), and the 8 avoidance items (scoring range:0-40).
Change from 1 month Generic health-related quality of life related to gynaecological cancer at 12 months post RT/RTBT | 12 months
  Generic health-related quality of life (QoL) related to gynaecological cancer is assessed with the Dutch version of the European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire Core 30 (QLQ-C30). The QLQ-C30 is composed of 5 functional scales (resp. physical, role, cognitive, emotional, and social functioning) and 9 symptom scales and/or items (fatigue, nausea and vomiting, pain, dyspnoea, insomnia, appetite loss, constipation, diarrhoea, and financial difficulties), and a global health status/QoL scale. All scales/item measures have scoring ranges from 0-100. A high scale score for a functional scale represents a high/healthy level of functioning. A high scale score for a symptom scale/item scale represents a high level of symptomatology/problems. A high scale score for the global health status/QoL represents high QoL. For scoring principles, please see the EORTC QLQ-C30 Scoring Manual.
change from 1 month in Psychological distress at 12 months post RT/RTBT | 12 months
  Psychological distress is assessed with the Dutch version of the 14-item Hospital Anxiety and Depression Scale (HADS). The HADS consists of two 7-item subscales, measuring anxiety (scoring range: 0-21) and depression (scoring range: 0-21). Higher scores on subscales indicate higher levels of anxiety and/or depression. (measured at 1, 3, 6, 12 months post RT/RTBT).
Change from 1 month in Relationship dissatisfaction at 12 months post RT/RTBT | 12 months
  Relationship dissatisfaction is assessed with the 10-item relationship dissatisfaction subscale of the Maudsley Marital Questionnaire (MMQ; scoring range 0-80). Higher scores represent greater dissatisfaction. (measured at 1, 3, 6, 12 months post RT/RTBT).
Change from 1 month in Frequency of dilator use at 12 months post RTBT | 12 months
  Patients treated with RTBT will in addition complete questions regarding the frequency of dilator use during the previous month. (measured at 1, 3, 6, 12 months post RTBT).
Change from baseline in Vaginal symptoms at 12 months post RT/RTBT | 12 months
  Vaginal symptoms will be assessed during physical examination. Vaginal symptoms include grade of mucosal atrophy, dryness, fibrosis, and signs of vaginal shortening and/or stenosis. Vaginal symptoms will be recorded using the Common Terminology Criteria for Adverse Events (CTCAE) v.4.037. (measured at 1, 3, 6, 12 months post RT/RTBT).
Cost-effectiveness | 12 months
  A cost-effectiveness analysis will be conducted in which the costs of the intervention will be related to shifts in other health care costs and the impact on patient outcome. A cost-price analysis will be performed for the nurse-led intervention (including training, counselling hours and materials). Other health care use will be limited to sexuality-related health care utilization (including gynaecologist, radiation oncologist, general practitioner, psychologist, and sexologist), estimated from patient reports and valued using standard prices. the Dutch tariff for the EuroQol 5 Dimensions 5 Levels (EQ-5D-5L) will be used (measured at 1, 3, 6, 12 months post RT/RTBT).

OTHER OUTCOMES:
Treatment credibility and expectancy for improvement | at 1 month post RT/RTBT
  Treatment credibility and expectancy for improvement will be assessed using the 4-item Credibility and Expectancy Questionnaire (CEQ; scoring range: 4-36). Higher scores indicate higher expectations of the intervention (for intervention group) or care as usual (for control group).

CONTACTS AND LOCATIONS:
Overall Officials: Moniek M ter Kuile, PhD, Study Chair — Leiden University Medical Center; Carien L Creutzberg, MD, PhD, Principal Investigator — Leiden University Medical Center; Jan Willem M Mens, MD, Principal Investigator — Erasmus Medical Center
Locations (8):
- Netherlands (8):
  - Academic Medical Center, Amsterdam
  - Radiotherapiegroep, Arnhem
  - Catharina Hospital, Eindhoven
  - University Medical Center Groningen, Groningen
  - MAASTRO clinic, Maastricht
  - Radboudumc, Nijmegen
  - Erasmus MC, Rotterdam
  - University Medical Center Utrecht, Utrecht

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bakker RM, ter Kuile MM, Vermeer WM, Nout RA, Mens JW, van Doorn LC, de Kroon CD, Hompus WC, Braat C, Creutzberg CL. Sexual rehabilitation after pelvic radiotherapy and vaginal dilator use: consensus using the Delphi method. Int J Gynecol Cancer. 2014 Oct;24(8):1499-506. doi: 10.1097/IGC.0000000000000253. PMID 25248115
- [Background] Bakker RM, Mens JW, de Groot HE, Tuijnman-Raasveld CC, Braat C, Hompus WC, Poelman JG, Laman MS, Velema LA, de Kroon CD, van Doorn HC, Creutzberg CL, Ter Kuile MM. A nurse-led sexual rehabilitation intervention after radiotherapy for gynecological cancer. Support Care Cancer. 2017 Mar;25(3):729-737. doi: 10.1007/s00520-016-3453-2. Epub 2016 Oct 27. PMID 27787681
- [Background] Bakker RM, Vermeer WM, Creutzberg CL, Mens JW, Nout RA, Ter Kuile MM. Qualitative accounts of patients' determinants of vaginal dilator use after pelvic radiotherapy. J Sex Med. 2015 Mar;12(3):764-73. doi: 10.1111/jsm.12776. Epub 2014 Nov 25. PMID 25424559
- [Background] Vermeer WM, Bakker RM, Stiggelbout AM, Creutzberg CL, Kenter GG, ter Kuile MM. Psychosexual support for gynecological cancer survivors: professionals' current practices and need for assistance. Support Care Cancer. 2015 Mar;23(3):831-9. doi: 10.1007/s00520-014-2433-7. Epub 2014 Sep 14. PMID 25218609
- [Derived] Suvaal I, Hummel SB, Mens JM, Tuijnman-Raasveld CC, Tsonaka R, Velema LA, Westerveld H, Cnossen JS, Snyers A, Jurgenliemk-Schulz IM, Lutgens LCHW, Beukema JC, Haverkort MAD, Nowee ME, Nout RA, de Kroon CD, van den Hout WB, Creutzberg CL, van Doorn HC, Ter Kuile MM. Efficacy of a nurse-led sexual rehabilitation intervention for women with gynaecological cancers receiving radiotherapy: results of a randomised trial. Br J Cancer. 2024 Sep;131(5):808-819. doi: 10.1038/s41416-024-02775-8. Epub 2024 Jul 3. PMID 38961193
- [Derived] Suvaal I, Hummel SB, Mens JM, van Doorn HC, van den Hout WB, Creutzberg CL, Ter Kuile MM. A sexual rehabilitation intervention for women with gynaecological cancer receiving radiotherapy (SPARC study): design of a multicentre randomized controlled trial. BMC Cancer. 2021 Dec 4;21(1):1295. doi: 10.1186/s12885-021-08991-2. PMID 34863145